CLINICAL TRIAL: NCT06879067
Title: A Phase I Study of the Safety, Tolerability and Immune Effects of the Nasal Anti-CD3 Monoclonal Antibody Foralumab in Healthy Human Volunteers
Brief Title: Safety, Tolerability and Immune Effects of the Nasal Foralumab in Healthy Human Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tiziana Life Sciences LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: 134155
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Safety; Tolerability
Keywords: foralumab; safety; tolerability; phase 1

STUDY DESIGN:
Intervention Model Description: This is a randomized, double blind Phase I dose escalation study evaluating three dose levels of Foralumab via intranasal administration from single-dose vials. Each dose group will complete 7 days of assessment and be evaluated for safety before the study moves to the next dosing level. After the first 9 subjects complete their Day 8 visit, the next 9 subjects will be enrolled and receive 50 ug of nasal Foralumab or placebo once daily for 5 days; after the second group completes visit Day 8, the third dose group will be enrolled and receive 250 ug of nasal Foralumab/placebo once daily for 5 days.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The treating physician and subjects will be blinded to treatment. The BWH IDS pharmacy will have the treatment code assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- nasal foralumab 10 μg daily (Experimental): Group A: nasal foralumab 10 μg daily for 5 days
  Interventions: Drug: Foralumab Nasal
- nasal foralumab 50 μg daily (Experimental): Group B: nasal foralumab 50 μg daily for 5 days
  Interventions: Drug: Foralumab Nasal
- nasal foralumab 250 μg daily (Experimental): Group C: nasal foralumab 250 μg daily for 5 days
  Interventions: Drug: Foralumab Nasal
- placebo (Placebo Comparator): The placebo was acetate buffer. It was handled in a manner identical to active drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo nasal spray
  Arms: placebo
Drug: Foralumab Nasal — foralumab nasal spray
  Arms: nasal foralumab 10 μg daily; nasal foralumab 250 μg daily; nasal foralumab 50 μg daily

SUMMARY:
The goal is to establish the safety of administration of nasal foralumab to healthy volunteers in escalating doses to determine the dose at which immune effects are observed. Patients will receive doses for 5 consecutive days and have a follow-up period.

DETAILED DESCRIPTION:
This was a randomized, double blind phase 1 dose escalation study evaluating 3 dose levels of foralumab via intranasal administration from single-dose vials. The rationale behind the proposed research was to establish an immunologically active dose of foralumab given by the nasal route. Given that foralumab has never been administered by the nasal route to humans, this was a safety and dose finding study. Each dose group was observed until Day 7 to assess safety before moving to the next higher dose. This study also helped determine the dose at which immune effects (induction of regulatory T cells and changes in cytokine profiles of immune cells) were observed in subjects treated with foralumab.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ages 18 to 65 years
* Healthy adults
* Ability and willingness to provide informed consent and comply with study requirements and procedures

Exclusion Criteria:

* Chronic medical disease compromising organ function
* Corticosteroids within the past month
* Pregnancy or lactating
* Inflammatory bowel disease, rheumatoid arthritis, systemic lupus erythematosus, asthma, thyroid disease, or type I diabetes
* Chronic rhinitis, deviated septum, nasal polyps, history of sinusitis treated within the past year.
* Participation in another clinical trial within the past 30 days
* Known history of drug or ETOH abuse
* Screening labs outside of the normal range; EBV IgM positive subjects with clinical signs will not receive study drug
* Nasal corticosteroids; antihistamines; nasal flu dosing within 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2020-11-09 (Actual)

PRIMARY OUTCOMES:
Safety- Adverse Events | Day 1 vs End of Study (Day 30)
  Establish the safety of administration of nasal Foralumab to healthy volunteers in escalating doses for 5 consecutive days. Two or more serious adverse events occur that are possibly, probably or definitely related to nasal Foralumab.
Immune Effect | Dat 1 vs End of Study (Day 30)
  Determine the dose at which immune effects are observed in subjects treated with Foralumab

CONTACTS AND LOCATIONS:
Locations (1):
- Ann Romney Center for Neurologic Diseases, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No